CLINICAL TRIAL: NCT05881226
Title: Application of Biomarkers in Neurological Diseases
Status: Recruiting | Type: Observational
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: Bio-Neuro
Record Dates: First submitted 2023-05-15; First posted 2023-05-31 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to hospital/emergency department with neurological diseases: All clinical data, laboratory data and imaging data of patients at baseline and follow-up were collected, as well as blood and tissue samples that did not affect the diagnosis and treatment of patients after obtaining the consent of patients at different time points in the acute and chronic phases.

SUMMARY:
To explore the predictive and diagnostic role of biomarkers in patients with neurological diseases.

DETAILED DESCRIPTION:
With the rise and continuous development of omics technology and bioinformatics technology, some scholars have applied proteomics technology and metabolomics technology to study the brain tissue, plasma and CSF of patients with nervous system diseases, so as to screen out potential biomarkers, with a view to providing new research ideas for pathogenesis and early diagnosis of neurological diseases. At present, the research on some novel biomarkers is still in its infancy, and many key problems remain to be solved. It is necessary to further determine the expression level of biomarkers in normal human body and the characteristics of biomarkers in patients with neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with neurological diseases;
2. Subjects or legal agents agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Participating in other clinical investigators;
2. Unwilling to be followed up or poor treatment compliance;
3. Other conditions considered unsuitable for inclusion by the researchers.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with neurological diseases admitted to hospital/emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
mRS score in 90 days | 3 months
  The proportion of 3-month good functional outcome (mRS Score 0-2) in patients with neurological diseases was evaluated by mRS Score

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China